CLINICAL TRIAL: NCT03883971
Title: Effects of 3D Printing Technology on Maternal Fetal Bonding Compared to 2D/3D Ultrasounds
Brief Title: Third Trimester 3D Printed Models Versus 3D Ultrasound Effects on Maternal-Fetal Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: John Cote (Unknown)
Responsible Party: Principal Investigator, Amy Badura Brack, Professor, Creighton University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1052761-4
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Maternal-Fetal Relations

STUDY DESIGN:
Intervention Model Description: 3D ultrasound only or 3D ultrasound and printed model of fetal face
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D model (Experimental): patient is given 3D printed model of her fetus's face
  Interventions: Other: 3D printed model
- picture (Placebo Comparator): patient is given a fetal picture only.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 3D printed model — Same as previously reported in arm descriptions
  Arms: 3D model
Other: Placebo — nothing other than the ultrasound
  Arms: picture

SUMMARY:
This study will invite healthy women with singleton pregnancies and normal 20 week ultrasounds to participate in the study that will involve completing a demographic questionnaire and measure of attachment, a 3D ultrasound, being randomized to receive a 3D printed model of the fetal face or not, and completing the attachment measure again.

ELIGIBILITY:
Inclusion Criteria:

* women
* between19-45 years of age
* singleton pregnancy
* no less than 26-weeks pregnant and no more than 31-weeks pregnant at randomization
* normal fetal anatomic survey (fas) ultrasound
* fluent in English

Exclusion Criteria:

* additional medical or entertainment ultrasounds after the 20 week anatomic ultrasound

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Singleton Pregnancy
Enrollment: 96 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Maternal Antenatal Attachment Scale (MAAS) | 5 minutes
  The MAAS is a 19 item questionnaire measuring maternal-fetal attachment. Each item has five answer choices scored from 1 low attachment to 5 high attachment such that the total score ranges from 19 to 95. The measure also includes two subscales: (1) Quality of Attachment has 10 items with a range of 10-50 and measures the quality of the mother's attachment to her fetus. (2) Time measures the time spent in attachment mode (or intensity of preoccupation) and consists of 8 items for a range of 8 to 40. (for clarity one item included in the total score is not included in either subscale.)

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton Univeristy, Omaha, Nebraska, United States